CLINICAL TRIAL: NCT05994105
Title: Integration of Augmented Reality in Expressive Art Therapy for Borderline Personality Features
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahria University (Other)
Responsible Party: Principal Investigator, Zohra Batool, PhD Scholar, Bahria University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Bahria University
Record Dates: First submitted 2022-11-18; First posted 2023-08-16 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Self Destructive Behavior; Mood Disturbance; Self Esteem
MeSH Terms: conditions — Self-Injurious Behavior | interventions — Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): individuals who will not receive the management plan
- Experimental Group (Experimental): Individuals who will receive therapy
  Interventions: Behavioral: Art based Augmented Reality

INTERVENTIONS:
Behavioral: Art based Augmented Reality — The participants will be provided 14 sessions management plan
  Other Names: Psychotherapy
  Arms: Experimental Group

SUMMARY:
From the last decades, applied approach for the use of augmented reality on clinical and health psychology has grown exponentially. Hence, the present study is aimed to examine the effectiveness of augmented reality for the treatment of borderline personality features in young adults. For the purpose, it is hypothesized that (i) borderline personality features of experimental groups will be reduced in posttest followed by the integration of augmented reality in expressive art therapy (ii) Borderline personality features of experimental group will decrease significantly as compared to control group in the post test followed by the integration of augmented reality in expressive art therapy (iii) Borderline personality feature of self-destruction will be reduced in posttest followed by the integration of augmented reality in expressive art therapy (iv) Borderline personality feature of affect regulation will be reduced in posttest followed by the integration of augmented reality in expressive art therapy and (v) Borderline personality feature of negative self-perception will be reduced in posttest followed by the integration of augmented reality in expressive art therapy. For the present purpose, a total of 20 subjects experiencing symptoms of Borderline personality features will be screened and recruited from the Umeed e Nau clinics of the Institute of Professional Psychology Bahria University Karachi Campus by initial screening of the subjects. Participants will be monitored through pre and post-screening of Borderline Symptoms Checklist assigned to an experimental (treatment group) and control (waiting list) group using convenient sampling. The experimental group will receive the Management plan; which will be comprised of total 14 sessions. The effectiveness of the intervention plan will be measured via quantitative measure (the latest version of SPSS).

DETAILED DESCRIPTION:
The final sample consisted of 20 participants (aged 18-36, males n=5, and females n=15). Half of the sample was assigned to the intervention group, while the other half was assigned to the control group as per convenient sampling method. The intervention group participants were provided with a total of fourteen psychotherapy sessions at Umeed-e-Nau clinic at the Institute of Professional Psychology.

Assemblr Studio: Easy AR Maker (android version 4.1.7) Assemblr studio was used to make augmented reality within the sessions. It is a free android application for turning 2-D and 3-D images into augmented reality. The application was designed by Assemblr (2018) and consists of a marker less based type of augmentation. Rather it uses basic templates and camera picture upload options, transforming a simple image into augmented reality format. It also provides drag and drop options and does not require any coding.

3-D Pen/ Doodling pen A digital 3-D pen was used to contrast art in the sessions. It was a portable and handheld type of machine.

Procedure Approval to conduct this research was taken from the board of the Institute of Professional Psychology, Bahria University, Karachi Campus. The participants were then approached via advertisement on social media platforms highlighting awareness regarding borderline personality features and the objectives of the present research. The sample frame consisted of 36 individuals which were then screened for the inclusion criteria using the Borderline symptoms list. The final 20 participants were then randomly divided into two equal groups, namely the treatment group and the control waiting-list group. The final 20 participants were all made privy to the details and purpose of the research and their consent was taken. Confidentiality was maintained and the participants retained the right to withdraw their participation at any point in the study, as well as remain able to decide not share details of specific traumatic or hurtful life events. Moreover, the researchers took all necessary steps to ensure safety of the participants' wellbeing.

The experimental group's treatment plan for augmented reality-based art therapy interventions comprised of 14 weekly individual standard sessions. Each session was of approximately 90 minutes, duration of which was divided into 5 minutes initial check-in to reflect participant's outer world, 30 minutes for making art, 30 minutes for discussing the art, 10 minutes to wrap up the session, and 5 minutes final check-out to reflect on the session's interventions, explorations, and learning.

The treatment plan was divided into three levels. Level one comprised of three primary intervention-based sessions designed to help build rapport and have the participants get familiar with intervention's concept. Level two, lasting from session four to session twelve, dealt with gradually evolving the participants' perceptual continuum to a developmental continuum where the individual would the be able to make desired changes and recreate their thoughts, feelings, and behaviors. The third and final level included sessions thirteen, fourteen, and the consequent follow-ups. Its purpose was to reflect upon the participants' learning so far and to sum up the termination phase of therapy. The follow-up session took place three weeks after the unilateral termination of the regular sessions. Here the participants were required to complete the Borderline Symptoms List (Bohus et al., 2007), and if it was assessed that a participant needed further therapeutic help, they were provided with referrals to professionals. The control group participants were also assessed for post-test borderline symptoms at this point of time.

After the completion of the study, the results were coded and analyzed using SPSS version 22.0.

Session Plan Session 01 - GROW (The Kitchen Table Classroom, 2019). The aim of this session was to develop rapport with the participant through semi structured interview and goal setting. The objective of the session was to explore the concept of personal change in clients via art medium where they drew the word GROW and self-reflected from their onwards.

Session 02 - Scribble zoom in and out (Khat & Macklin, 2019). The aim of the session was to facilitate the process of catharsis, and have the client engage in and explore their impulsivity and curiosity. Moreover, childhood insecurities and traumas were explored in this session as well and the artwork was used to discuss the participant's self-perception of change.

Session 03 - Blind Contour Drawing (Hu et al., 2021). The aim of the session was to psychoeducate the participant with the primary goal of using blind contour drawing to draw attention towards differences of perceptions and conceptualization of information. The objective of this intervention was to help the participant become aware of their own judgmental reactions in different life circumstances.

Session 04 - Self-Awareness via Johari's window (Batool, 2018). The aim of the session was to introduce the concept of thought modification via developing insight through blind spots, in a nonjudgmental and nonthreatening manner. The objective of the session's activity was to help the participant become self-aware and to bring positive change in self-development.

Session 05 - My Life Outline (Batool, 2018). The aim of the session was to address self-harming behavior in session by identifying distressing elements in the participant's life, and to learn to better cope with these distressing elements in a nonjudgmental manner. The objective was to have the participant become able to identify different distressing and pleasant moments in their life, eventually leading to development of insight and stability in mood regulation.

Session 06 - Free Flow Writings without stimulus (Batool, 2018). The aim of the session was to channel emotional distress, negative thoughts, and self-destructive behavior. It was based upon the presumption that, while everybody has something to say and the ability to say it, the mental wellspring may be blocked by apathy, self-criticism, resentment, anxiety about deadlines, fear of failure or censure, or other forms of resistance. Objective was to explore and discuss features of personality malfunctions.

Session 07 - Draw what you hear (Chowdhury, 2019). The aim of the session was to provide the participant with cathartic medium to anchor their self, with respect to emotional distress and mood regulation. The objective was that via this integration of the self, the participant would then be able to regulate their free affirmative emotions.

Session 08 - Draw your breath (Batool, 2018). The aim of the session was to strengthen self-awareness, which eventually helped the participant to maintain mood, regulate self-image, and possibly reduce self-harm. Objective was to help the participant feel relief by the end of the session.

Session 09 - Body Healing in Ink (Batool, 2018). The aim of the session was to reduce the participant's aggressive and suicidal impulses, thus, helping them better cope with their self-destructive behavior. In this manner, the objective of the session was to utilize and project participant's aggression in making art in a nonjudgmental manner.

Session 10 - Paint inside a Heart (Khat & Macklin, 2019). The aim of the session was to provide the participant with a nonthreatening and nonjudgmental medium through which they may process the emotions being experienced in that moment. The objective of the session was to bring into awareness the participant's own emotional burdens and help them create a positive self-image.

Session 11 - Sculpture of Anger (Godfrey, 2008). The aim of the session was to have the participant become aware of their emotional distress and the ways in which they manage that distress. To attain this goal, the participant was asked to create an art form sculpture that most resembled their anger in real life. By the end of session, the participant was then able to become self-aware of their aggression and frustration, which automatically led to a reduction in tendency to self-harm and helped them better regulate their mood.

Session 12 - Words of Mind Haiku (Stephenson & Rosen, 2015). The aim of the session was to provide the participant with a unique way to become mindful of their progress, enabling them to manage their borderline personality features in healthy way. The objective of the session was to have the participant self-reflect and then accept their self-image. By the end of the session, the participant was able to write their creative thoughts in form of poems, helping them to understand compassion and self-regulation.

Session 13 - Recollection of Moments (Filmore, 2019). The aim of the session was to reflect upon the growth and improvement observed by the participant as well as the therapist. In the session, progress exhibited by the participant was discussed and goals of the therapy process were reviewed. At last, one final objective was to ready the participant for termination of therapy.

Session 14 - What I Have. Aim of the session was to talk about the developmental continuum of the participant, to explore their awareness and acceptance of recreational thoughts while taking examples from their real-life scenarios. Therapy was terminated and closure was provided.

Follow-up session. It took place three weeks after the termination session. In the follow-up session, the participants completed formal post-Intervention assessment of the Borderline Symptoms List (Bohus et al, 2007). Moreover, if required, further referrals and psychiatric consultations were made for the participant with their agreement.

Statistical Analysis The pre- and post-intervention assessments of the treatment group and the control group for the Borderline Symptoms List (Bohus et al., 2007) was scored. The results were coded and exported to SPSS, version 22.0. The data was then analyzed with paired sample analysis to explore the possible significant differences between scores of BSL of treatment group as compared to control group.

ELIGIBILITY:
Inclusion Criteria

* Age comprises of young adults above 18 years (minimum) to 36 years (maximum) with at least academic qualification of 12th grade.
* Individuals whose raw score on elation (50 or above) or percentile 50 or above on a scale of Borderline Symptoms Checklist in pre assessment phase.
* Participants who subjectively rate on 50 or above on personal state of borderline symptoms checklist.
* Participants who has no prior record of diagnosis of Borderline personality disorder.
* Participants who were not go into psychological consultations (past or present).
* Participants who were not go into psychiatric consultations (past or present).
* Individuals who were ready to volunteer, committed and motivated to undertake the interventions.
* Individuals who thinks that face instant Interpersonal conflicts (Pseudo or Meta conflict).
* Individuals who believe that their daily living is unable to bear for them (suicidal ideation).
* Participants who has social support at present (both through informal networks (social mediums and in person).
* Participants who understand the language instruction of i.e. Basic English and Urdu language.
* Willing to agree for in-person therapy. Exclusion Criteria
* History of physical illness or organic brain damage; especially in the last few years.
* Any related medication taken or medication being taken now in this regard.
* Age of young adults below 18 years to and above 36 years.
* Individuals who raw score on low (49 or below) or percentile 49 or below on a scale of Borderline Symptoms Checklist in pre assessment phase.
* Participants who subjectively rate on 49 or below on personal state of borderline symptoms checklist.
* Participants who has a prior record of diagnosis of Borderline personality disorder.
* Active or recent physical addiction to alcohol or drugs.
* Individuals with already receiving psychological therapy or psychiatric consultations for the same matter.
* Individuals who are involved in persistent suicide risk who require proper health management.
* Participants who opt for online therapy.

Ages: 19 Years to 36 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-11-12 (Actual)

PRIMARY OUTCOMES:
Borderline Symptoms Checklist | four months
  The Borderline Symptoms List (Bohus et al, 2007) was used as self-report measure to assess the participants' level of borderline personality features. It is comprised of 95 total items which are rated using a 5-point Likert scale where 0 = not at all and 4 = very strongly. The test is reported to have internal consistency Cronbach's α = 0.97. Moreover, BSL has seven subscales, namely, self-perception, affect regulation, dysphoria, loneliness, intrusions, hostility, and the self-destruction subscale which measures aspects of suicidal ideation, self-harm behavior, longing for death, and fascination with death using 12 items with a Cronbach's α = 0.94.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Professional Psychology, Bahria University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No